CLINICAL TRIAL: NCT06932887
Title: Mountain West Arthritis Secondary Prevention Program - The Beat Pain Better Trial
Brief Title: The Beat Pain Better Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Julie Fritz, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00182708; 1U48DP006833 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis; Chronic Pain Management
Keywords: osteoarthritis; chronic pain; physical therapy; self-management
MeSH Terms: conditions — Osteoarthritis; Chronic Pain | interventions — methyl hydroxyethyl cellulose

STUDY DESIGN:
Intervention Model Description: This trial uses a multiple randomization design. There are two randomizations; one to a text messaging strategy. The second randomization for those who enroll is to a Walk with Ease format.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Text Messaging (Active Comparator): Weekly text message invitations over 4 weeks to engage in physical activity counseling
  Interventions: Behavioral: Text Messaging
- Text Messaging with Motivational Messages (Experimental): Weekly text message invitations over 4 weeks to engage in physical activity counseling that also include motivational messages
  Interventions: Behavioral: Text Messaging; Behavioral: Motivational Messaging
- PA Counseling and Self-Directed Walk with Ease (Active Comparator): Six weeks of weekly telehealth PA counseling provided by a physical therapist plus connection to the Walk with Ease portal for ongoing self-management.
  Interventions: Behavioral: Physical Activity Counseling and Self-Directed Walk with Ease
- PA Counseling and Enhanced, Self-Directed Walk with Ease (Experimental): Six weeks of weekly telehealth PA counseling provided by a physical therapist plus connection to the Walk with Ease portal for ongoing self-management along with opportunity to participate in group classes.
  Interventions: Behavioral: Physical Activity Counseling and Self-Directed Walk with Ease; Behavioral: Enhanced Walk with Ease

INTERVENTIONS:
Behavioral: Text Messaging — Weekly SMS messages sent to potential participants to inform them of the opportunity to participate in PA counseling for their arthritis. instructions also provided on how to request a referral.
  Arms: Text Messaging; Text Messaging with Motivational Messages
Behavioral: Motivational Messaging — The use of short motivational messages along with text messages inviting persons to participate in PA counseling. The messages are intended to enhance the motivation to participate in PA counseling.
  Arms: Text Messaging with Motivational Messages
Behavioral: Physical Activity Counseling and Self-Directed Walk with Ease — All persons consenting to PA counseling receive 6 weekly sessions provided in-person or remote with 2-way video or audio commu¬nication. All participants receive education to address negative psy-chological appraisals of OA, reassur¬ance that PA is safe and beneficial, and a PA program primarily focused on walk¬ing, although additional activities may be included. Additional components include exercises tai¬lored to the partici¬pant's needs and coping strategies such as mindful breathing to help manage stress.
  Arms: PA Counseling and Enhanced, Self-Directed Walk with Ease; PA Counseling and Self-Directed Walk with Ease
Behavioral: Enhanced Walk with Ease — Along with the portal registration participants in the Enhanced WWE group are also offered the opportunity to participate in virtual group WWE classes offered on a rolling basis in either English or Spanish.
  Arms: PA Counseling and Enhanced, Self-Directed Walk with Ease

SUMMARY:
The Beat Pain Better study examines strategies to increase the reach of evidence-based interventions for persons with osteoarthritis (OA) in communities that experience disparities. The study is a hybrid type 3 effectiveness-imple-mentation trial using sequential, multiple assignment, ran¬domi¬zation to evaluate 1) two text mes¬saging strat¬egies to reach persons with OA and enroll them in physical activity counseling provided by physical therapists; and 2) two strat¬egies to engage enrolled persons in the Walk with Ease (WWE) intervention for sustained self-management.

DETAILED DESCRIPTION:
We will conduct a hybrid type 3 effectiveness-imple¬mentation trial with a sequential, multiple assignment, ran¬domi¬zed design. Primary outcome is physical activity (PA) counseling reach (Aim 1). Secondary outcomes evaluate reach of WWE (Aim 2) and outcomes across RE-AIM domains (Aim 3). Persons with ICD-10 diagnosis codes indicating OA will be identified from EHRs in partnering clinics and sent text message (TM) invitations to participate in PA counseling. Phase I randomization will test two TM strategies: weekly TMs over 4 weeks with or without motiva¬tional messages. Phase II randomization for those who enroll in PA counseling and provide consent will test two formats for the WWE AAEBI; self-directed or enhanced self-directed delivery.

Participants will be randomized with 1:1 distribution at each randomization. Participants may consent and enroll for randomization to a WWE format even if they did not receive the TM intervention. The first randomization is performed using the TM platform (Azara or similar), stratified by site. The second randomization is performed using the REDCap randomization module, also stratified by site and by baseline PA level. Randomization schemas will be developed before enrollment. Randomization errors will be recorded as protocol deviations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45 or older;
2. Visit in participating medical clinic within the past 6 months
3. OA diagnosis code related to lower extremity and/or spine on the problem list or associ¬ated with an encounter in the past 6 months
4. Has functioning cell phone able to receive calls and texts

Exclusion Criteria:

1. Unable to participate in a regular walking program defined as the ability to walk for at least five minutes with or without the use of an assistive device.
2. Medical contraindication to participation in physical activity
3. Unable to communicate in either Spanish or English

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 346 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Reach-Enroll for PA Counseling | From time of initiating text messaging to enrollment
  Number of persons enrolling in PA counseling divided by the total number of persons eligible for enrollment

SECONDARY OUTCOMES:
PEG-3 | Baseline, 6, 12 and 26 weeks
  The PEG-3 is a self-report measure that includes 3 items evaluating 1) pain severity; and interference of pain with 2) enjoyment and 3) general activity. Item response options range from 0-10. The PEG-3 score is expressed as the mean of all item scores ranging from 0-10
PROMIS Physical Function | Baseline, 6, 12 and 26 weeks
  The PROMIS short form 6b for physical function is a self-report that uses fixed items from the PROMIS physical function item bank to provide a T-score with population mean = 50 (sd=10).
PROMIS Sleep Disturbance | Baseline, 6, 12 and 26 weeks
  The PROMIS short form 6a for sleep disturbance is a self-report that uses fixed items from the PROMIS sleep disturbance item bank to provide a T-score with population mean = 50 (sd=10).
PROMIS Depression | Baseline, 6, 12 and 26 weeks
  The PROMIS short form 8a for depression is a self-report that uses fixed items from the PROMIS depression item bank to provide a T-score with population mean = 50 (sd=10).
Sleep Duration | Baseline, 6, 12 and 26 weeks
  The Sleep Duration Question asks; "During the past month, how many hours and minutes of actual sleep did you get at night?" Response is recorded in hours and minutes
Pain Self-Efficacy | Baseline, 6, 12 and 26 weeks
  The Pain Self-Efficacy Scale is a 4-item scale assessing a person's confidence of persons to achieve goals and perform activities even with pain. Each item is scored from 0-6 for an overall score ranging from 0-24.
High Impact Chronic Pain | 6, 12 and 26 weeks
  High impact chronic pain is based on responses to two questions; "In the past 3 months, how often do you have pain?" and "Over the past 3 months, how often did pain limit your life or work activities?" Response options for both questions are (0) Never, (1) Some Days, (2) Most days, (3) Every Day. A score of 2 or 3 on BOTH questions indicates the person has HICP.
Physical Activity | Baseline, 6, 12 and 26 weeks
  The physical activity questionnaire asks respondents about their participation in physical activity and exercise within the past 6 weeks in 6 categories: 1) light physical activity (such as laundry, vacuuming, making beds or dusting); 2) moderate physical activity (such as scrubbing floors, washing windows, gardening or raking leaves); 3) heavy physical activity (such as carrying heavy objects, heavy digging, pushing a mower or hard manual labor); 4) light physical exercise (such as leisurely walking or slow dancing); 5) moderate physical exercise (such as hiking or swimming); and 6) vigorous physical exercise (such as jogging or playing tennis singles). For each category that the respondent indicates participating in, an additional question asks about the frequency at which they carried out these activities: ≤1 time/month, 2-3 times/month, 1-2 times/week, 3-4 times/week, 5-6 times/week, or daily
Global Impression of Change | 6, 12 and 26 weeks
  Participants are asked their overall level of satisfaction with treatment with responses on a likert scale.
Health care utilization | 6, 12 and 26 weeks
  Self-reported utilization of surgery, injections, imaging or other discrete interventions for pain associated with arthritis

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Utah, Salt Lake City, Utah
  - Association for Utah Community Health, Salt Lake City, Utah
  - Vamos Health, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in a data repository
Supporting Information: Study Protocol, SAP